CLINICAL TRIAL: NCT00332709
Title: An Open Phase III Trial With Letrozole Alone or in Combination With Zoledronic Acid as Extended Adjuvant Treatment of Postmenopausal Patients With Primary Breast Cancer
Brief Title: Safety/Efficacy of Letrozole Monotherapy or in Combination With Zoledronic Acid as Extended Adjuvant Treatment of Postmenopausal Patients With Primary Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345DDE09
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Results first posted 2011-11-16 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-10

CONDITIONS: Osteoporosis; Postmenopausal
Keywords: Breast cancer; postmenopausal; bone mineral density; Zoledronic acid; Letrozole; extended adjuvant treatment.; Postmenopausal women with primary hormone receptor positive breast cancer
MeSH Terms: conditions — Osteoporosis; Breast Neoplasms | interventions — Letrozole; Zoledronic Acid

ARMS (2):
- Letrozole (Experimental): Letrozole orally 2.5 mg/day for 3 years
  Interventions: Drug: Letrozole
- Letrozole + Zoledronic Acid (Experimental): Letrozole orally 2.5mg/day for 3 years; Zoledronic acid 4mg every 6 months by infusion
  Interventions: Drug: Letrozole; Drug: Zoledronic acid

INTERVENTIONS:
Drug: Letrozole — 2.5 mg/day for 3 years
Drug: Zoledronic acid — 4 mg every 6 months
  Arms: Letrozole + Zoledronic Acid

SUMMARY:
This was a prospective, randomized, open-label, two arm phase III trial designed to evaluate the efficacy and safety of zoledronic acid in preventing bone loss in postmenopausal women with operable breast cancer who had received 4 to 6 years of adjuvant tamoxifen therapy after resection of the tumor. Patients were treated with letrozole 2.5 mg orally per day or letrozole 2.5 mg orally per day in combination with zoledronic acid 4 mg/6 months as an infusion.

This trial did not recruit patients in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Compliant postmenopausal women with primary operable breast cancer after 4 to 6 years of therapy with tamoxifen (end of tamoxifen therapy within last 6 months)
* Performance status 0-2 (Eastern Cooperative Oncology Group)
* Patients without severe osteoporosis at study entry
* No evidence of relapse at the time of randomization
* Adequate function of bone marrow, kidney, and liver

Exclusion Criteria:

* Estrogen- and progesterone-receptor status negative or unknown
* Completion of adjuvant tamoxifen therapy more than 6 months prior to study start
* Inflammatory breast cancer
* Current/active dental problems including infection of the teeth or jawbone, dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw, of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery
* History of diseases with influence on bone metabolism such as Paget's disease and primary overactive parathyroid
* Prior or concomitant therapies: chemotherapy within the last 12 months, intravenous or oral bisphosphonates, systemic corticosteroids, anabolic steroids or growth hormones, Tibolone, parathyroid hormone, systemic sodium fluoride or any drugs known to affect the skeleton (such as calcitonin, mithramycin, or gallium nitrate)
* Patients with previous or concomitant cancers (not breast cancer) within the past 5 years EXCEPT adequately treated basal or squamous cell skin cancers or in situ cancer of the cervix. Patients with previous other cancer(s) must have been disease-free for at least 5 years.
* Patients currently receiving oral bisphosphonates must discontinue these at least 3 weeks prior to study start.

Additional protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2006-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- Germany (23):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Deggendorf
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Georgsmarienhütte
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Halle
  - Novaertis Investigative Site, Hamein
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Höxter
  - Novartis Investigative Site, Ilsede
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Leer
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Salzgitter
  - Novartis Investigative Site, Schwenningen
  - Novartis Investigative Site, Stendal
  - Novartis Investigative Site, Völklingen
  - Novartis Investigative Site, Witten

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total Randomized participants were 83. 2 patients were enrolled but never received study medication. Hence, 81 were included in the safety population.
Groups:
- Letrozole: Letrozole 2.5 mg/day for 3 years
- Letrozole + Zoledronic Acid: Letrozole 2.5mg/day for 3 years plus Zoledronic acid 4mg every 6 months
Period: Overall Study
Arm/Group | Letrozole | Letrozole + Zoledronic Acid
Started | 40 | 41
Completed | 24 | 21
Not Completed | 16 | 20
Not completed — Adverse Event | 11 | 14
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Administrative Problems | 0 | 3
Not completed — Abnormal test procedure result | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Letrozole + Zoledronic Acid | Total
Number analyzed (Participants) | 37 | 39 | 76
Age, Categorical [Count of Participants; unit: Participants] — Demographic data is provided for the Intent to Treat population.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 37 | 39 | 76
    >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 61.3 (7.3) | 58.4 (7.3) | 59.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 39 | 76
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density (BMD) From Baseline to Month 36
Description: Change in bone mineral density (BMD) measured by dual X-ray absorptiometry (DXA) in lumbar spine (L1-L4). Change calculated by (Month 36 BMD-Baseline BMD)/Baseline BMD*100.
Time Frame: at 36 months as compared to baseline
Population: (ITT) The study population will consist of post menopausal breast cancer patients who have completed 4 to 6 years of adjuvant Tamoxifen therapy after therapy. Participants with observations at both baseline and endpoint were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Letrozole | Letrozole + Zoledronic Acid
Number analyzed (Participants) | 21 | 20
Percent | -0.11 (0.14) | 0.03 (0.08)

2. Secondary Outcome: Change in Bone Mineral Density From Baseline to 12 Months
Description: as for outcome 1
Time Frame: Baseline, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Letrozole | Letrozole + Zoledronic Acid
Number analyzed (Participants) | 23 | 23
g/cm^2 | -0.04 (0.04) | 0.02 (0.05)

3. Secondary Outcome: Number of Participants With Any Kind of Fractures, by Visit.
Description: Number of participants with fractures of any type since the last visit
Time Frame: Baseline, Month 6, 12, 18, 24 , 30 and 36
Population: (ITT) The study population will consist of post menopausal breast cancer patients who have completed 4 to 6 years of adjuvant Tamoxifen therapy after therapy. Participants with observations from baseline to month 36 were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Letrozole | Letrozole + Zoledronic Acid
Number analyzed (Participants) | 21 | 20
Participants
  Baseline | 0 | 0
  Month 6 | 0 | 0
  Month 12 | 0 | 0
  Month 18 | 0 | 0
  Month 24 | 0 | 0
  Month 30 | 0 | 0
  Month 36 | 0 | 0

4. Secondary Outcome: Median Disease Free Survival (DFS)
Description: Disease Free Survival is measured in days and represents the number of days participants were progression free. Progression free survival is defined as the time from randomization to the date of the first documented progression or recurrence of disease or death from any cause. Median disease free survival is the time when 50% of the patients had a recurrence.
Time Frame: 36 months
Population: (ITT) The study population will consist of post menopausal breast cancer patients who have completed 4 to 6 years of adjuvant Tamoxifen therapy after therapy. The median disease free survival was not observed because patients in the combination therapy did not have any recurrences.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Letrozole | Letrozole + Zoledronic Acid
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Percent Change in Bone Mineral Density (BMD) From Baseline to Month 36
Description: Bone Mineral Density is measured by dual energy x-ray absorptiometry (DXA) scan.
  ANCOVA model was used in the analysis where: Variable = Baseline, Center, Treatment BMD = (Month 36 BMD-Baseline BMD)/Baseline BMD*100.
Time Frame: Baseline, Month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change in BMD
Arm/Group | Letrozole | Letrozole + Zoledronic Acid
Number analyzed (Participants) | 21 | 20
Percent Change in BMD | -11.34 (17.72) | 3.31 (8.32)

6. Primary Outcome: Change in T-score From Baseline to Month 36
Description: BMD measured by DXA (dual energy x-ray absorptiometry) at lumbar spine, L1-L4. The T-Score is a comparison of a patient's BMD to that of a healthy 30 year of the same sex and ethnicity. The criteria of the World Health Organization are Normal is a T-Score of 1.0 or higher. Osteopenia is defined as between - 1.0 and -2.5. Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and half standard deviations below the mean of a 30 year old man/woman.
Time Frame: Baseline and Month 36
Population: (ITT) The study population will consist of post menopausal breast cancer patients who have completed 4 to 6 years of adjuvant Tamoxifen therapy after therapy.Participants with observations at both baseline and endpoint were included in the analysis.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Letrozole | Letrozole + Zoledronic Acid
Number analyzed (Participants) | 20 | 21
T-Score | -0.90 (1.03) | 0.46 (0.27)

7. Primary Outcome: Change in Z Score From Baseline to Month 36
Description: Bone Mineral Density is measured by dual energy x-ray absorptiometry (DXA). The Z-Score is the number of standard deviations a patient's BMD differs from the average BMD of their age, sex and ethnicity. A Z-score of less than minus -1.5 raises concern of factors other than aging as contributing to osteoporosis.
Time Frame: Baseline, month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Letrozole | Letrozole + Zoledronic Acid
Number analyzed (Participants) | 22 | 20
Z-Score | -0.31 (0.35) | 0.25 (0.34)

8. Secondary Outcome: Change in T-Score From Baseline to Month 12
Description: as for outcome 6
Time Frame: Baseline, Month 12
Population: (ITT) The study population will consist of post menopausal breast cancer patients who have completed 4 to 6 years of adjuvant Tamoxifen therapy after therapy. Participants with observations at both baseline and endpoint were included in this analysis.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Letrozole | Letrozole + Zoledronic Acid
Number analyzed (Participants) | 23 | 24
T-Score | -0.31 (0.35) | 0.25 (0.34)

9. Secondary Outcome: Change in Z-Score From Baseline to Month 12
Description: (DXA). The Z-Score is the number of standard deviations a patient's BMD differs from the average BMD of their age, sex and ethnicity. A Z-score of less than minus -1.5 raises concern of factors other than aging as contributing to osteoporosis
Time Frame: Baseline, Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Letrozole | Letrozole + Zoledronic Acid
Number analyzed (Participants) | 23 | 22
Z-Score | -0.26 (0.35) | 0.37 (0.38)

ADVERSE EVENTS:
Groups:
- Letrozole + Zolendronic Acid: Letrozole 2.5mg/day for 3 years plus Zoledronic acid 4mg every 6 months
Arm/Group | Letrozole | Letrozole + Zolendronic Acid
Serious Adverse Events (participants affected / at risk) | 6/40 | 7/41
Other Adverse Events (participants affected / at risk) | 35/40 | 35/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=40) | Letrozole + Zolendronic Acid (N=41)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 1 | 0
CONCOMITANT DISEASE PROGRESSION (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 | 1
OXYGEN SATURATION DECREASED (Investigations) | 0 | 1
AXILLARY MASS (Musculoskeletal and connective tissue disorders) | 1 | 0
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=40) | Letrozole + Zolendronic Acid (N=41)
VERTIGO (Ear and labyrinth disorders) | 2 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 4
CONSTIPATION (Gastrointestinal disorders) | 3 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 3
DRY MOUTH (Gastrointestinal disorders) | 3 | 3
DYSPEPSIA (Gastrointestinal disorders) | 2 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 7
CHILLS (General disorders) | 1 | 7
FATIGUE (General disorders) | 2 | 12
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 3
OEDEMA PERIPHERAL (General disorders) | 4 | 3
PYREXIA (General disorders) | 0 | 9
HEPATIC CYST (Hepatobiliary disorders) | 3 | 0
CYSTITIS (Infections and infestations) | 2 | 0
NASOPHARYNGITIS (Infections and infestations) | 3 | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 11 | 14
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 5
BONE PAIN (Musculoskeletal and connective tissue disorders) | 12 | 14
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 6
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 5
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 1
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 5 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 10
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 0
HEADACHE (Nervous system disorders) | 5 | 9
MIGRAINE (Nervous system disorders) | 2 | 1
DEPRESSION (Psychiatric disorders) | 2 | 1
SLEEP DISORDER (Psychiatric disorders) | 2 | 3
ATROPHIC VULVOVAGINITIS (Reproductive system and breast disorders) | 3 | 0
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 2 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 4
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 | 6
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 3
HOT FLUSH (Vascular disorders) | 9 | 9
LYMPHOEDEMA (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or disclosure of the trial results in their entirety.